CLINICAL TRIAL: NCT01153477
Title: Effectiveness of an Enhanced Adaptive Continuing Care Model for Cocaine Dependence
Brief Title: Effectiveness of Enhanced Treatments for Drug Dependence
Acronym: EETDD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 810112
Record Dates: First submitted 2010-06-24; First posted 2010-06-30 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAU (No Intervention): This group is the control group by which we are comparing our intervention. This group will not receive an intervention from us but will continue to be treated at the Intensive Outpatient facility from which we recruited them.
- Counseling (TMAC-E) (Experimental): This telephone based intervention includes six factors to improve our extended treatment model: Incentive component; Patient choice; Provision of cell phones to those who need them; Social support and community resources; Positive recovery factors; and Outreach following dropout.
  Interventions: Behavioral: Telephone Monitoring and Counseling - Enhanced

INTERVENTIONS:
Behavioral: Telephone Monitoring and Counseling - Enhanced — Calls or in-person sessions, 1x weekly for first 8 weeks, then every other week up to a year. Step up session frequency if needed based on participants' ratio of protective and risk factors.
  Arms: Counseling (TMAC-E)

SUMMARY:
The purpose of this challenge grant is to conduct an initial test of a new, enhanced version of this protocol (telephone monitoring and counseling - enhanced, or TMAC-E), which has been modified to include the elements of our existing continuing care intervention plus patient-centered changes to boost patient involvement and community linkages. The investigators will recruit 150 cocaine dependent patients in publicly funded, community-based programs and randomize them to treatment as usual or the TMAC-E and follow them for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* (1) qualify for a DSM-IV diagnosis of cocaine dependence, with some cocaine use in the prior 6 months;
* (2) be 18 to 75 years of age;
* (3) have no current psychotic disorder or evidence of dementia severe enough to prevent participation in outpatient treatment;
* (4) have no acute medical problem requiring immediate inpatient treatment;
* (5) not be in methadone or other modes of Drug and Alcohol treatment, other than Intensive Outpatient Program;
* (6) be willing to be randomized and participate in research;
* (7) because of study follow-up requirements, subjects will be able to provide the name, verified telephone number, and address of at least one contact who can provide locator information on the patient during follow-up. We will include patients with dependence on other substances, provided that they are cocaine dependent and meet other inclusion criteria.

Exclusion Criteria:

* have a current psychotic disorder or evidence of dementia severe enough to prevent participation in outpatient treatment;
* have acute medical problem requiring immediate inpatient treatment;
* are in methadone or other modes of DA treatment, other than IOP;
* or cannot provide names of people who can get messages to them for follow up, in the event we cannot locate the participant at their original address and number. Also, if they are court mandated to treatment or otherwise considered a prisoner, they will be ineligible for the study as we have not applied for Subpart C approval.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Time Line Follow Back | 3 month
  abstinence from drug and alcohol use within each 3 month period of the follow-up (as indicated by the TLFB)
Time Line Follow Back | 6 month
  abstinence from drug and alcohol use within each 3 month period of the follow-up (as indicated by the TLFB)
Time Line Follow Back | 9 month
  abstinence from drug and alcohol use within each 3 month period of the follow-up (as indicated by the TLFB)
Time Line Follow Back | 12 month
  abstinence from drug and alcohol use within each 3 month period of the follow-up (as indicated by the TLFB)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States